CLINICAL TRIAL: NCT07038993
Title: Role of Venous Pressure Monitoring As a Predictor Of High-Flow Access In Prevalent Hemodialysis Patients
Brief Title: Venous Pressure Monitoring As a Predictor Of High-Flow Access In Prevalent Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ashraf Hassan, Lecturer of Internal Medicine and Nephrology, Faculty of Medicine, Ain shams University, Cairo, Egypt., Ain Shams University
Other Study IDs: FMASU MD221/2017
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Venous Pressure; Predictor; High Flow Access; Hemodialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Chronic hemodialysis patients of both sexes with autogenous arteriovenous fistulas.
  Interventions: Other: Venous Pressure Monitoring; Other: Color Doppler Ultrasound

INTERVENTIONS:
Other: Venous Pressure Monitoring — Measurement of venous pressure will be taken at dialysis machine pump speed set at 200ml/min, fistula needle gauge 16.
Other: Color Doppler Ultrasound — Arteriovenous fistula (AVF) Access flow (QA) will be obtained using color Doppler ultrasound using the Mindray-M5 ultrasound system. AVF feeding arterial flow will be measured immediately proximal to the fistula. The QA volume will be obtained using the algorithm available on the system, which is based on the mean flow of two measurements.

SUMMARY:
This study aimed to detect the possibility of using venous pressure as a predictor for high flow access as a simple, non-invasive screening technique in hemodialysis patients.

DETAILED DESCRIPTION:
The patient's vascular access is often referred to as their "lifeline," and without it, the life-sustaining treatment of hemodialysis would not be possible. To maintain access, patency depends on accurate diagnosis and timely, active interventions.

The Kidney Disease Outcomes Quality Initiative (K/DOQI) recommends native arteriovenous fistula (AVF) as the vascular access of choice for hemodialysis due to its longevity, lower complications, and lower mortality rate compared to catheters.

Currently, K/DOQI guidelines suggest that high intra-access pressure may be regarded as a surrogate for arteriovenous fistula (AVF) outflow stenosis. It can be measured using static venous pressure (sVP) or standardized dynamic venous pressure (dVP).

ELIGIBILITY:
Inclusion Criteria:

* Age from 28 to 81.
* Both sexes.
* Patients with the presence of an autogenous arteriovenous fistula (AVF) and a minimum hemodialysis treatment duration of six months.

Exclusion Criteria:

* Physical examination revealed signs of AVF outflow stenosis, including localized edema, collateral circulation, hyperpulsatile fistula characteristics, or a positive hand elevation test.
* If ultrasound confirmed AVF stenosis or thrombosis, or angiography identified central venous stenosis or thrombosis in clinically suspected cases.

Ages: 28 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective cohort study enrolled 59 chronic hemodialysis patients of both sexes with autogenous arteriovenous fistula (AVF).
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Static venous pressure | 6 months post-procedure
  Static venous pressure (SVP) were measured with the blood pump deactivated through direct intra-access measurement via the venous outflow cannulation needle. Blood pressure (BP)-adjusted values were calculated using the patient's mean arterial blood pressure (MAP) recorded contemporaneously with venous pressure measurements.

SECONDARY OUTCOMES:
Standardized dynamic venous pressure | 6 months post-procedure
  Standardized dynamic venous pressure (sDVP) measurements were performed with the hemodialysis machine blood pump calibrated to deliver 200 ml/min within five minutes of treatment initiation, utilizing a standardized 16-gauge venous outflow cannulation needle for measurement consistency.
Arteriovenous fistula flow | 6 months post-procedure
  Arteriovenous fistula flow (Qa) was quantified using a Mindray-M5 US system with integrated flow calculation algorithms. Feeding arterial blood velocity and vessel diameter measurements were obtained approximately 2 cm proximal to the fistula anastomosis. Flow calculations were based on the mean of two independent measurements, and patients demonstrating US evidence of stenosis or thrombosis were excluded from further analysis.
Urea reduction ratio | 30 minutes following treatment completion
  Urea reduction ratio (URR) was subsequently calculated as an indicator of hemodialysis treatment adequacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.